CLINICAL TRIAL: NCT02966197
Title: the Efficacy of Prophylactic Internal Iliac Artery Balloon Catheterization in the Management of Placenta Previa and Accreta
Brief Title: Efficacy of Prophylactic Internal Iliac Artery Balloon Catheterization in the Management of Placenta Previa and Accreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deng Dongrui (Other)
Responsible Party: Sponsor-Investigator, Deng Dongrui, professor, chief doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-C20150516
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Placenta Previa; Placenta Accreta
MeSH Terms: conditions — Placenta Previa; Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon group (Experimental): Prophylactic Internal Iliac Artery Balloon Catheterization
  Interventions: Procedure: prophylactic internal iliac artery balloon catheterization; Device: Prophylactic internal iliac artery balloon; Radiation: Radiology operation
- Control group (No Intervention): no intervention

INTERVENTIONS:
Procedure: prophylactic internal iliac artery balloon catheterization — Between June 2015 and August 2016
  Arms: Balloon group
Device: Prophylactic internal iliac artery balloon
  Arms: Balloon group
Radiation: Radiology operation
  Arms: Balloon group

SUMMARY:
Placenta previa and accreta both could potentially cause serious postpartum hemorrhage and even maternal death. Interventional radiological techniques have been developed to limit massive hemorrhage during caesarean section. This study investigated the efficacy of prophylactic internal iliac artery balloon catheterization in management for placenta previa and accreta.

DETAILED DESCRIPTION:
Placenta previa and accreta both could potentially cause serious postpartum hemorrhage and even maternal death. Interventional radiological techniques have been developed to limit massive hemorrhage during caesarean section. This study investigated the efficacy of prophylactic internal iliac artery balloon catheterization in management for placenta previa and accreta. Between June 2015 and August 2016,patients were personally recruited and managed by the authors,and assigned to either balloon group or control group by their willingness to catheterization or not. Both groups benefitted similar management protocol with the exception of interventional radiology operation. Intraoperative blood loss, transfusion volume, radiation dose, exposure time, surgical duration, procedure complications and neonatal outcomes were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women were eligible if they were diagnosed to have placenta previa and accreta by sonographic examination or Magnetic Resonance Imaging.

Exclusion Criteria:

* Any case who had bleeding disorder or underwent emergency cesarean delivery was excluded.

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
blood loss | intraoperative

SECONDARY OUTCOMES:
operation duration | intraoperative
fluid transfusion | intraoperative
blood transfusion | intraoperative

IPD SHARING:
Plan to Share IPD: Undecided